CLINICAL TRIAL: NCT02698228
Title: Regional Anaesthesia for Painful Injuries After Disasters (RAPID) Study: A Randomized Trial
Brief Title: Regional Anaesthesia for Painful Injuries After Disasters
Acronym: RAPID
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study did not occur
Sponsor: Epicentre (Other)
Collaborators: Brown University (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Epicentre RAPID Trial
Record Dates: First submitted 2016-02-16; First posted 2016-03-03 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Lower Limb Injuries; Fracture
Keywords: anesthesia
MeSH Terms: conditions — Fractures, Bone | interventions — Bupivacaine; Morphine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care (Sham Comparator): Intravenous injection of 0.1mg/kg of morphine. Injection of 5cc of 0.9% normal saline into the subcutaneous tissue of the thigh.
  Interventions: Drug: Morphine
- Femoral nerve block (Active Comparator): Intravenous injection of 0.1mg/kg of morphine. Injection of 20cc of 0.5% bupivacaine into the fascia iliaca space using standard anatomic landmarks.
  Interventions: Drug: Bupivacaine (femoral nerve block); Drug: Morphine
- Ultra-sound guided femoral nerve block (Active Comparator): Intravenous injection of 0.1mg/kg of morphine.Injection of 20cc of 0.5% bupivacaine around their femoral nerve under direct ultrasound guidance
  Interventions: Drug: Bupivacaine (femoral nerve block); Drug: Morphine; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacaine (femoral nerve block) — 0.5% bupivacaine
  Arms: Femoral nerve block; Ultra-sound guided femoral nerve block
Drug: Morphine — Intravenous injection of 0.1mg/kg of morphine
Device: Ultrasound
  Arms: Ultra-sound guided femoral nerve block

SUMMARY:
The goal of the RAPID study is to fundamentally transform the way serious injuries are managed after earthquakes and other disasters by introducing a novel and cost-effective method for pain control. The study will enroll patients in the aftermath of a major earthquake to determine whether regional anesthesia, either with or without ultrasound-guidance, can reduce suffering from lower limb injuries, the most common earthquake-related injury, above and beyond the current standard of care for pain control in these settings.

DETAILED DESCRIPTION:
The Regional Anaesthesia for Painful Injuries after Disasters (RAPID) study aims to evaluate whether regional anesthesia (RA), either with or without ultrasound (US) guidance, can reduce pain from earthquake-related lower limb injuries in a disaster setting. The proposed study is a blinded, randomized controlled trial among earthquake victims with serious lower extremity injuries in a resource-limited setting. After obtaining informed consent, study participants will be randomized in a 1:1:1 allocation to either: standard care (parenteral morphine at 0.1 mg/kg); standard care plus a landmark-guided fascia iliaca compartment block (FICB); or standard care plus an US-guided femoral nerve block. General practice humanitarian response providers who have undergone a focused training in RA will perform nerve blocks with 20 ml of 0.5% levobupivacaine. US sham activities will be used in the standard care and FICB arms and a normal saline injection will be given to the control group to blind both participants and non-research team providers. The primary outcome measure will be the summed pain intensity difference calculated using a standard 11-point numerical rating scale reported by patients over 24-hours of follow-up. Secondary outcome measures will include overall analgesic requirements, adverse events and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) presenting to an MSF field hospital with one or more lower limb injuries .

Exclusion Criteria:

* multi-system trauma
* severe respiratory distress
* hypotension
* altered mental status
* active infection at the sight of injection
* known current pregnancy
* unable to provide informed consent.
* known allergies to local anesthetic agents or narcotic pain medication
* receiving antithrombotic therapy or with a preexisting coagulopathy
* likely to receive regional anesthesia for alternative reasons within two hours of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 24 hours
  The summed pain intensity difference (SPID), a widely used measure for assessing the efficacy of new methods for pain management will be administered before and 24 hours for all patients.

SECONDARY OUTCOMES:
Analgesic requirements | 24 hours
  Analgesic requirements will be recorded as the total amount of analgesic medication received during the full 24 hours of patient follow up.
Patient satisfaction | 24 hours
  All patients will be assessed at 24 hours for their overall satisfaction with their pain management on a standard Likert scale
Serious Adverse Events | 24 hours
  The investigators will monitor all patients for serious adverse events, including allergic reaction or local anesthetic systemic toxicity (LAST) from the regional anesthesia or respiratory depression or hypotension from narcotic pain medications

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca F Grais, PhD, Study Director — Epicentre

IPD SHARING:
Plan to Share IPD: Yes
The trial dataset will be made publicly available at the conclusion of the trial.

REFERENCES:
- [Derived] Levine AC, Teicher C, Aluisio AR, Wiskel T, Valles P, Trelles M, Glavis-Bloom J, Grais RF. Regional Anesthesia for Painful Injuries after Disasters (RAPID): study protocol for a randomized controlled trial. Trials. 2016 Nov 14;17(1):542. doi: 10.1186/s13063-016-1671-z. PMID 27842565